CLINICAL TRIAL: NCT00283465
Title: An Open-label, Randomized Study to Evaluate the Effect of Early Treatment of Anemia With Epoetin Alfa on Hemoglobin, the Incidence of Blood Transfusions and Quality of Life in Patients Receiving Platinum-containing Chemotherapy
Brief Title: A Study of the Effectiveness and Safety of Treatment With Epoetin Alfa on Hemoglobin Levels, Red Blood Cell Transfusions, and Quality of Life in Patients With Cancer Receiving Platinum-containing Chemotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag B.V. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR002047
Record Dates: First submitted 2006-01-27; First posted 2006-01-30 (Estimated); Last update posted 2011-01-14 (Estimated); Status verified 2011-01

CONDITIONS: Anemia; Neoplasm
Keywords: Anemia; cancer; neoplasm; transfusion; quality of life; tumor response; survival; chemotherapy; hemoglobin; standard care; epoetin alfa; epoetin; erythropoietin
MeSH Terms: conditions — Anemia; Neoplasms | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: Epoetin alfa

SUMMARY:
The purpose of this study is to compare the effectiveness of early treatment of anemia with epoetin alfa (a glycoprotein that stimulates red blood cell production) or best standard anemia care on the need for blood transfusions, tumor response, anemia and quality of life in patients with cancer receiving platinum-containing chemotherapy.

DETAILED DESCRIPTION:
Cancer patients often experience anemia due to the disease itself, chemotherapy, or both. Quality of life is also affected, due in part to the tiredness associated with anemia. Previous studies with epoetin alfa have suggested that epoetin alfa increases hemoglobin and reduces the incidence of red blood cell transfusions and that achieving a higher hemoglobin level may improve quality of life. This is a randomized, open-label, multicenter study that evaluates the effects of early treatment with epoetin alfa compared with standard anemia care alone to determine its impact on the need for blood transfusions, tumor response, anemia and quality of life, as well as on the safety of epoetin alfa when used in the prevention of anemia during chemotherapy in adult patients with cancer. Patients will receive epoetin alfa injections (10,000 units) under the skin 3 times a week until 4 weeks after the last day of the last chemotherapy cycle, in addition to best standard care, or best standard care alone. Best standard care during chemotherapy may include red blood cell transfusions, white cell growth factors, and iron supplementation, as needed. The dose of epoetin alfa may be adjusted up (to 20,000 units) or down (to 75% of the last dose) based on hemoglobin level.

The primary measure of effectiveness will be determined by the number of patients who receive an allogenic red blood cell transfusion during the study and during each chemotherapy cycle. Additional measures of effectiveness include: the average number of units transfused during each cycle, change in quality of life (feeling of well-being, as assessed by responses to 3 different patient questionnaires), change in hemoglobin level, relationship between change in hemoglobin and quality of life, tumor response, and the number of patients surviving up to 12 months after the end of treatment. Safety evaluations (incidence of adverse events, clinical laboratory tests, vital signs, and physical examinations) will be performed throughout the study. The study hypothesis is that treatment with epoetin alfa will reduce the need for red blood cell transfusions, increase hemoglobin levels, improve quality of life, and result in a positive tumor response in patients with cancer who are receiving chemotherapy. This study will be conducted in the Netherlands and will only enroll European patients. Patients will receive epoetin alfa injections (10,000 units) under the skin 3 times a week until 4 weeks after the last day of the last chemotherapy cycle, or best standard care. Dose may be adjusted up (to 20,000 units) or down (to 75% of the last dose) based on hemoglobin level.

ELIGIBILITY:
Inclusion Criteria:

* Patients having a confirmed diagnosis of cancer and are planned to receive platinum chemotherapy with a minimum of 8 weeks on study and a maximum of 6 or 12 cycles
* Eastern Cooperative Oncology Group (a scale used by researchers to represent the level of activity that a patient is capable of) score of 0 (able to carry out all normal activity without restriction) to 3 (capable of only limited self-care, confined to bed or chair >50% of waking hours)
* life expectancy of >=5 months
* have a hemoglobin value of <=7.5 grams per deciliter at any time during or prior to chemotherapy

Exclusion Criteria:

* Patients having clinically significant disease/dysfunction of the pulmonary, cardiovascular, endocrine, neurological, gastrointestinal, or genitourinary systems that is not due to cancer or chemotherapy (this disease/dysfunction is only an exclusion criterion if it causes an expected early withdrawal from the study)
* uncontrolled high blood pressure
* history of seizures
* untreated iron, folate, or vitamin B12 deficiency
* received androgen (e.g., testosterone) therapy within 2 months of study entry, had a major illness within 7 days of study entry, or a major infection within 1 month of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 1999-11; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Number of patients who receive an allogenic red blood cell transfusion during the study, during each chemotherapy cycle, and at 4 weeks after the last administration of chemotherapy

SECONDARY OUTCOMES:
Number of units transfused during each chemotherapy cycle; change in quality of life; change in hemoglobin level; relationship between change in hemoglobin and quality of life; tumor response; patient survival up to 12 months after the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag B.V. Clinical Trial, Study Director — Janssen-Cilag B.V.

REFERENCES:
- [Result] Savonije JH, van Groeningen CJ, van Bochove A, Honkoop AH, van Felius CL, Wormhoudt LW, Giaccone G. Effects of early intervention with epoetin alfa on transfusion requirement, hemoglobin level and survival during platinum-based chemotherapy: Results of a multicenter randomised controlled trial. Eur J Cancer. 2005 Jul;41(11):1560-9. doi: 10.1016/j.ejca.2005.03.024. PMID 15953714